CLINICAL TRIAL: NCT00733044
Title: Cost-effectiveness of Multidisciplinary Management of Tinnitus at a Specialised Tinnitus Centre
Brief Title: Cost-effectiveness of Multidisciplinary Management of Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Iris Maes, MSc, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 06-0012; ZonMw 80-007022-98-07715
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Tinnitus
Keywords: Objective tinnitus; Tinnitus; RCT; Specialised treatment; Usual care; Cost-effectiveness
MeSH Terms: conditions — Tinnitus | interventions — Patient Care Team

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialized Care (Experimental): Stepped-care cognitive behavioural approach with elements from tinnitus retraining therapy
  Interventions: Behavioral: Specialized Care
- Usual Care (Active Comparator): Audiological diagnostics and intervention and, if necessary, one or more consultations with a social worker with a maximum of ten one hour session
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Specialized Care — The intervention consists of the integration of integral tinnitus management provided by a specialized tinnitus centre in the health care system. The tinnitus centre offers care following a stepped-care approach with two levels. The first level of intervention consists of audiological diagnostics and intervention, a tinnitus educational group session and a individual consult with a clinical psychologist. For patients with mild complaints this basic intervention is expected to suffice. For patients with moderate to severe complaints a second level of intervention exists. This level of intervention consists of combinations of the following therapies: Cognitive Behavioural Therapy (CBT), Attention Diversion (AD), exposure techniques, and Relaxation Therapy (RT).
  Other Names: Multidisciplinary care
  Arms: Specialized Care
Other: Usual Care — Usual care consists of a standardized version of treatment that is currently applied in peripheral audiological centres throughout the Netherlands. A telephone survey was conducted amongst all audiological centres (n=28) in the Netherlands. The results of this survey determined the content of the usual care treatment protocol in the current study. The treatment consists of audiological diagnostics and intervention and, if necessary, one or more consults with a social worker with a maximum of ten one hour sessions.
  Arms: Usual Care

SUMMARY:
Background: Tinnitus is a common chronic health condition that affects 10% to 20% of the general population. Among severe sufferers it causes disability in various areas. As a result of the tinnitus quality of life is often impaired. At present there is no cure or uniformly effective treatment, leading to fragmentized and costly tinnitus care. Evidence suggests an integral multidisciplinary approach in treating tinnitus is effective. The main objective of this study is to examine the effectiveness, costs, and cost-effectiveness of an integral treatment provided by a specialized tinnitus center versus usual care. This paper describes the study protocol.

Methods/Design: In a randomized controlled clinical trial 198 tinnitus patients will be randomly assigned to a specialized tinnitus care group or a usual care group. Adult tinnitus sufferers referred to the audiological centre are eligible. Included patients will be followed for 12 months.

Primary outcome measure is generic quality of life (measured with the Health Utilities Index Mark III). Secondary outcomes are severity of tinnitus, general distress, tinnitus cognitions, tinnitus specific fear, and costs. Based on health state utility outcome data the number of patients to include is 198. Economic evaluation will be from a societal perspective.

Discussion/ Conclusion: This is, to our knowledge, the first randomized controlled trial that evaluates an integral treatment of tinnitus that includes a full economic evaluation from a societal perspective. If this intervention proves to be effective and cost-effective, implementation of this intervention is considered and anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Subjective tinnitus complaints
* Referred to Tinnitus centre Limburg

Exclusion Criteria:

* Not being able to write and read in Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2007-09; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Generic Quality of Life as measured with the Health Utilities Index Mark 3 (HUI3) | At baseline and 3, 8 and 12 months follow-up

SECONDARY OUTCOMES:
Tinnitus related disability and handicap as measured with the Tinnitus Handicap Inventory (THI) | At baseline and at 3, 8 and 12 months follow-up
Tinnitus annoyance and severity, as measured with the Tinnitus Questionnaire (TQ) | At baseline and at 3, 8 and 12 months follow-up
Tinnitus-related fear was assessed by the Fear of Tinnitus Questionnaire (FTQ) | At baseline and at 3, 8 and 12 months follow-up
Dysfunctional beliefs and/or cognitions regarding the tinnitus, as measured with the Tinnitus Coping and Cognition list (TCCL) | At baseline and at 3, 8 and 12 months follow-up
Catastrophic (mis)interpretations of tinnitus, as measured with the Tinnitus Catastrophising Scale (TCS). | At baseline and at 3, 8 and 12 months follow-up
Costs, as measured with a retrospective cost questionnaire | At baseline and at 3,8 and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Johan WS Vlaeyen, Prof, PhD, Principal Investigator — Maastricht University; Manuela A Joore, PhD, Principal Investigator — Maastricht University Medical Center; Lucien J Anteunis, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Hoensbroeck Audiological Centre, Hoensbroek, Limburg, Netherlands

REFERENCES:
- [Derived] Cima RF, Maes IH, Joore MA, Scheyen DJ, El Refaie A, Baguley DM, Anteunis LJ, van Breukelen GJ, Vlaeyen JW. Specialised treatment based on cognitive behaviour therapy versus usual care for tinnitus: a randomised controlled trial. Lancet. 2012 May 26;379(9830):1951-9. doi: 10.1016/S0140-6736(12)60469-3. PMID 22633033
- [Derived] Cima R, Joore M, Maes I, Scheyen D, Refaie AE, Baguley DM, Vlaeyen JW, Anteunis L. Cost-effectiveness of multidisciplinary management of Tinnitus at a specialized Tinnitus centre. BMC Health Serv Res. 2009 Feb 11;9:29. doi: 10.1186/1472-6963-9-29. PMID 19210767